CLINICAL TRIAL: NCT02764658
Title: Studies in Pulmonary Inflammation and the Effectiveness of Pulmonary Recovery in COPD Patients：the Mechanism of Proteoglycan 4
Brief Title: Proteoglycan 4 Mechanism the Effectiveness of Pulmaonry Recovery in COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Shu-Chuan Ho, School of Respiratory Therapy, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: TMU-JIRB Ho1.2/20160212
Record Dates: First submitted 2016-05-01; First posted 2016-05-06 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ventilators, Negative-Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pulmonary recovery on the AECOPD (Experimental): Study in the pulmonary inflammation and the effectiveness of pulmonary recovery in AECOPD Patients
  Interventions: Device: Pulmonary recovery on the AECOPD; Other: Routine care on the AECOPD; Other: Routine care on the stable COPD
- Routine care on the AECOPD (Other): Study in the pulmonary inflammation and the effectiveness of pulmonary recovery in AECOPD Patients
  Interventions: Other: Routine care on the AECOPD; Other: Routine care on the stable COPD
- Routine care on the stable COPD (Other): Study in the pulmonary inflammation and the effectiveness of pulmonary recovery in stabel COPD Patients
  Interventions: Other: Routine care on the stable COPD

INTERVENTIONS:
Device: Pulmonary recovery on the AECOPD — The combination effect of negative pressure ventilation, limb muscle exercise training program and fibit monitor on acute exacerbation of AECOPD. To investigate the daily physical activity in routine care patients with after AECOPD and stable stage.
  Other Names: Ergometer for limb muscle training; Negative pressure ventilator; Fibit monitor
  Arms: Pulmonary recovery on the AECOPD
Other: Routine care on the AECOPD — To investigate whether daily physical activity、hypoxia and hyperinflation were associated with airway inflammation and PRG4 in Routine care patients wtih AECOPD and stable stage.
  Other Names: Physical daily activity; Fibit monitor
  Arms: Pulmonary recovery on the AECOPD; Routine care on the AECOPD
Other: Routine care on the stable COPD — To investigate whether daily physical activity、hypoxia and hyperinflation were associated with airway inflammation and PRG4 in Non-Pulmanary recovery patients wtih stable COPD.
  Other Names: Physical daily activity; Fibit monitor

SUMMARY:
The investigators previous research has demonstrated that proteoglycan 4 (PRG4) may be a biomarker for identification of severity in COPD. PRG4 was more sensitive and specific than CRP for confirming COPD severity and acute exacerbation frequency. It was related to the 1-year force vital capacity decline in COPD patients. The past study found that Prg4 is an immunomodulatory factor regulating parathyroid hormone actions on hematopoietic cells in mice. Previous report showed that voluntary wheel running and fluid flow shear stress that promote the expression of the Prg4 and association with pulmonary inflammation. COPD patients are characterized by a progressive decrease of lung function that is associated with increased in the airway and systemic inflammation. Pulmonary recovery (PR) is able to decrease acute exacerbation, maintain pulmonary function, increase exercise tolerance and improve quality of life in COPD patients, but it is unknown the mechanism of PRG4. The current study aimed to study in the pulmonary inflammation and the effectiveness of pulmonary recovery in COPD Patients：The mechanism of PRG 4.

DETAILED DESCRIPTION:
The investigators previous research has demonstrated that proteoglycan 4 (PRG4) may be a biomarker for identification of severity in COPD. PRG4 was more sensitive and specific than CRP for confirming COPD severity and acute exacerbation frequency. It was related to the 1-year force vital capacity decline in COPD patients. The past study found that Prg4 is an immunomodulatory factor regulating parathyroid hormone actions on hematopoietic cells in mice. Previous report showed that voluntary wheel running and fluid flow shear stress that promote the expression of the Prg4 and association with pulmonary inflammation. COPD patients are characterized by a progressive decrease of lung function that is associated with increased in the airway and systemic inflammation. Pulmonary recovery (PR) is able to decrease acute exacerbation, maintain pulmonary function, increase exercise tolerance and improve quality of life in COPD patients, but it is unknown the mechanism of PRG4. The current study aimed to study in the pulmonary inflammation and the effectiveness of pulmonary recovery in COPD Patients：The mechanism of PRG 4.

1. Proteoglycan 4 is correlated with pulmonary inflammation and decline of pulmonary function in the different phenotype of COPD.

   1-1 Classification of characteristic、the severity of disease、pulmonary functional test、exercise capacity and blood sample collection for routine analysis.

   1-2 Human blood bio-bank and molecular analysis: PRG4、IL-6、IL-8、TNFα、CRP& IL-10.

   1-3 To investigate whether daily physical activity、hypoxia and hyperinflation were associated with airway inflammation and PRG4 in COPD patients.
2. The mechanism of PRG 4 in the effectiveness of PR on the AECOPD. 2-1 The PR program: The combination effect of negative pressure ventilation and exercise training program on acute exacerbation of COPD (AECOPD).

   2-2 To examine the efficacy of PR on cytokines and PRG4 protein. 2-3 Correlation between PR effects and PRG4：PR is correlation with PRG4、clinical progression、exercise tolerance、PFT change and SpO2 during exercise.
3. In vitro cell culture research models 3-1 Pulmonary inflammatory model establishment：Human primary epithelium cell culture and Beas-2B for IL-1β、TNFα、LPS、IL-10 and H2O2 effects.

   3-2 Purification of peripheral blood monocyte cells：Primary culture to evaluate pulmonary inflammation and treatment effects.

   3-3 Hypoxia experiments：To test whether hypoxia induces regulation of PRG4 protein or different cytokines in epithelial cells.

   3-4 Inhibit PRG4：To prove the mechanism of PRG4 under the hypoxia model by PRG4 siRNA。
4. In vivo animal research models 4-1 Smoke-COPD mice models establishment： 4-2 To determinate the effects of exercise training in COPD mine. 4-3 To investigate on PRG4 protein in pulmonary inflammation and the effectiveness of exercise training in the tissue and serum of mice.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with acute exacerbation of COPD

  1. GOLD diagnostic criteria based on the COPD, the use of inhaled bronchodilators: the first second forced expiratory volume (FEV1.0) / forced vital capacity (FVC) <70%.
  2. Age ≧ 40 and ≦ 80 years old, is currently not accepting any research project.
  3. Physician assess the patient is currently in stable condition vital signs, complain dyspnea of exercise, consult RT for pulmonary rehabilitation.
  4. The purpose of this study by researchers explain, the researchers agreed to participate in this.

Stable COPD outpatients

1. GOLD diagnostic criteria based on the COPD, the use of inhaled bronchodilators: the first second forced expiratory volume (FEV1.0) / forced vital capacity (FVC) <70%.
2. Age ≧ 40 and ≦ 80 years old, is currently not accepting any research project.
3. The purpose of this study by researchers explain, the researchers agreed to participate in this.

Exclusion Criteria:

* Hospitalized patients with acute exacerbation of COPD

  1. Unstable vital signs: blood pressure <90 mm Hg, blood oxygen levels (SpO2) at Tx under still <85%.
  2. Associated with neuromuscular function disorders such as hemiplegia or no independent walking function.
  3. Have been diagnosed with severe mental disorders, such as dementia or or unable to cooperating people.

Stable COPD outpatients

1. Over the past three months there have been acute infection or are in a state of acute attacks.
2. Associated with neuromuscular function disorders such as hemiplegia or no independent walking function.
3. Have been diagnosed with severe mental disorders, such as dementia or unable to cooperating people

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
The systemic inflamation biomakers | 0~12 months
  Measured the proteaglycan4、IL-6、IL-8、TNFα、CRP& IL-10 from the supernatant with COPD patients

SECONDARY OUTCOMES:
Exercise capacity | 0~12 months
  Six-minute walking distance and lung
The correlaton with the exercise capacity and systemic inflammationcytokines | 0~12 months
  volumePulmonary recovery is correlation with PRG4、clinical progression、exercise tolerance、PFT change and SpO2 during exercise

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Chuan Ho, Principal Investigator — School of Respiratory Therapy, College of Medicine, Taipei Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ho SC, Lin HC, Kuo HP, Chen LF, Sheng TF, Jao WC, Wang CH, Lee KY. Exercise training with negative pressure ventilation improves exercise capacity in patients with severe restrictive lung disease: a prospective controlled study. Respir Res. 2013 Feb 19;14(1):22. doi: 10.1186/1465-9921-14-22. PMID 23421438
- [Background] Lee KY, Chuang HC, Chen TT, Liu WT, Su CL, Feng PH, Chiang LL, Bien MY, Ho SC. Proteoglycan 4 is a diagnostic biomarker for COPD. Int J Chron Obstruct Pulmon Dis. 2015 Sep 18;10:1999-2007. doi: 10.2147/COPD.S90926. eCollection 2015. PMID 26451097
- [Background] Wang CH, Chou PC, Joa WC, Chen LF, Sheng TF, Ho SC, Lin HC, Huang CD, Chung FT, Chung KF, Kuo HP. Mobile-phone-based home exercise training program decreases systemic inflammation in COPD: a pilot study. BMC Pulm Med. 2014 Aug 30;14:142. doi: 10.1186/1471-2466-14-142. PMID 25175787